CLINICAL TRIAL: NCT05113524
Title: The Effects of Dance on the Turning Characteristics of Patients With Parkinson's Disease During the Timed up and Go Test
Brief Title: Effects of Dance on the Turning Characteristics of Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: University of Wolverhampton (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Aline Nogueira Haas, Associate Professor, Federal University of Rio Grande do Sul
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 33547920.9.0000.5347; 12/18/NH/UOW (Registry Identifier: CAAE number)
Record Dates: First submitted 2021-10-28; First posted 2021-11-09 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Parkinson Disease(PD)
Keywords: Dance; Functional Mobility; Turning
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dance (Experimental): Dance intervention for 3 months, 2 times/week (1 instructor lecture session and 1 home session following a prepared video), 2 hours per week. Dance is a safe and effective form of activity, which has been used in PD population (Delabary et al., 2017; Sharp and Hewitt, 2014). Participants take part in a dance class specifically for people with PD lead by a qualified dance instructor. The dance class typically include a warm-up, dance related activities (specific to the genre of the class) and a cool-down.
  Interventions: Other: Dance
- Control Group (Active Comparator): Controls, not alter their personal lifestyle, but undergo the same testing as the exercise intervention group.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Dance — The dance program consists of 3 months of dance classes. Classes are specifically designed for people with Parkisnon's and lead by a qualified dance instructor experienced in teaching this population. The in-person dance classes are conducted in an appropriate room with chairs and ballet barres once a week. In addition, the participants received a CD containing a video of the recorded dance routine to be performed at home once a week. The class typically included a warm-up (10-15 min.), barre ballet exercises (10-15 min.), general dance-related activities (15-20 min), and a cool-down (10-15 min).
  Arms: Dance
Other: No intervention — Controls, not alter their personal lifestyle, but will undergo the same testing as the exercise intervention group.
  Arms: Control Group

SUMMARY:
The proposed control intervention trial, aims to analyse the effects of Dance in the turning characteristics in patients with Parkinson Disease (PD) using three- dimensional (3D) analysis during the timed up and go (TUG) test.

DETAILED DESCRIPTION:
Experimental Design: control intervention non-randomized trial. Search Location: University of Wolverhaptom, Walsall Campus, United Kingdom; Federal University of Rio Grande do Sul, Brazil.

Participants: 15 adults aged between 50 and 80 years, with a clinical diagnosis of idiopathic PD, staging between 1 and 4 of the Hoehn & Yahr Scale, recruited from Dance for Parkinson's Projects, West-Midlands County, United Kingdom, and from Parkinson's UK (United Kingdom).

Interventions: Dance intervention for 3 months, 2 times/week (1 instructor lecture session and 1 home session following a prepared video), 2 hours per week. Controls, not alter their personal lifestyle, but undergo the same testing as the exercise intervention group.

Outcomes: clinical-functional parameters (number of steps and total time of the 180 turning phase of the Timed up and go Test - TUG - and biomechanics parameter - girdle dissociation) Data Analysis: Data will be described by average values and standard deviation values. All statistical analyses will be carried out using SPSS version 23, and Microsoft Excel Program version 16.44. The significance level is set at p<0.05. The Cohen's d is going to be used to predict effect interpreted as small d= 0.2, medium d=0.5, and large d=0.8, and 95% confidence intervals were presented.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of PD according to the London Brain Bank Criteria;
* Able to understand the verbal instructions for the tests and to walk;
* Or attempt to walk independently with no walking aid.

Exclusion Criteria:

* Recent surgeries,
* Deep brain stimulation (DBS);
* Severe heart diseases, uncontrolled hypertension, myocardial infarction within a period of less than one year;
* Fitted with a pacemaker;
* Prostheses in the lower limbs;
* Stroke or other associated neurological diseases.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
180 turning phase of the Timed up and go Test (TUG) | Change from baseline at 3 months
  The beginning of the turning phase started from the last heel-strike of the regular straight line walking pattern. The end of the turn was the final heel-off at the end of the turning motion, where the participant was ambulating in the opposite direction and prior to the cyclic straight line gait pattern resuming. The exact time points were taken from the peak anterior-posterior linear velocity of the lower leg data corresponding with the specific heel-strike and heel-off instances. The number of steps and the total time taken to complete the 180 turning phase of the TUG test were measured.

SECONDARY OUTCOMES:
Girdle dissociation | Change from baseline at 3 months
  The girdle dissociation is a selected biomechanics parameter. To obtain the value for the girdle dissociation, the difference between the orientation of the pelvis and the affected shoulder in the transverse plane, was calculated for each data point throughout the 180 turning phase of the TUG test. The range between the maximum and minimum dissociation angles was reported and further analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Aline Nogueira Haas, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (2):
- Aline Nogueira Haas, Porto Alegre, Rio Grande do Sul, Brazil
- University of Wolverhampton, Walsall Campus, Walsall, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dos Santos Delabary M, Komeroski IG, Monteiro EP, Costa RR, Haas AN. Effects of dance practice on functional mobility, motor symptoms and quality of life in people with Parkinson's disease: a systematic review with meta-analysis. Aging Clin Exp Res. 2018 Jul;30(7):727-735. doi: 10.1007/s40520-017-0836-2. Epub 2017 Oct 4. PMID 28980176
- [Background] Dos Santos Delabary M, Monteiro EP, Donida RG, Wolffenbuttel M, Peyre-Tartaruga LA, Haas AN. Can Samba and Forro Brazilian rhythmic dance be more effective than walking in improving functional mobility and spatiotemporal gait parameters in patients with Parkinson's disease? BMC Neurol. 2020 Aug 18;20(1):305. doi: 10.1186/s12883-020-01878-y. PMID 32811464

DOCUMENTS (1):
  • Informed Consent Form (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT05113524/ICF_000.pdf